CLINICAL TRIAL: NCT05585697
Title: Markers of Bone Turnover and Advanced Glycation End Products Measured in the Circulation, Bone Marrow, and Bone Tissue in Individuals With and Without Type 2 Diabetes
Brief Title: Bone Turnover in Type 2 Diabetes and Non-diabetes Controls (DiaMarv)
Acronym: DiaMarv
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: AUH_HOK_2022_1
Record Dates: First submitted 2022-10-14; First posted 2022-10-19 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2; Bone Fragile
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood, bone marrow and bone tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 diabetes or control: Individuals with type 2 diabetes. Expect to include 26. Individuals without type 2 diabetes. Expect to include 26.
  Interventions: Other: None - crossectional

INTERVENTIONS:
Other: None - crossectional — None - crossectional

SUMMARY:
Type 2 diabetes (T2D) is related to an increased risk of major fractures which does written in English. The summary is used not only increase society health care costs, but also increase the morbidity and in the recruitment of peer reviewers.: mortality for patients with T2D. Traditional fracture predictors underestimate the risk in T2D. Thus, the bone affection is not caused by decreased bone mineral density but rather by impaired bone quality leading to fragile bone. In diabetes, circulating bone turnover markers are suppressed and advanced glycation endproducts may accumulate in the tissue. The study aims at exploring whether bone turnover in T2D is compromised in the circulation, bone marrow, and bone tissue and whether advanced glycation endproducts accumulate in these tissues. Furthermore, the investigators will assess whether bone turnover markers predict fractures in a cohort of individuals with diabetes. The project will contribute to the knowledge on bone disease in T2D and will ultimately benefit the patients by improving future fracture prevention strategies.

DETAILED DESCRIPTION:
3.1 Methods Study 1 is a cross-sectional study in which 26 individuals with T2D and 26 age matched individuals without T2D are examined. The investigators aim to investigate whether a) bone turnover markers are lower in individuals with type 2 diabetes (T2D) compared to persons without T2D based on circulating bone turnover markers, bone turnover markers in the bone marrow and bone turnover measured in bone tissue biopsies b) the levels of advanced glycation end-products (AGEs) in the circulation, bone marrow, bone tissue, and skin in individuals with and without T2D. The investigators hypothesize that the levels of AGEs is lower in all three tissue compartments in individuals with T2D compared to persons without T2D.

The individuals are included and recruited from outpatient clinics, general practitioners, letters based on information from national registries and via media advertisements.

Inclusion criteria for individuals with T2D; physician diagnosed T2D, diabetes duration ≥5 years, HbA1c ≥ 59 mmol/mol through the last 2 years, male gender, age > 40 years, and BMI < 35 kg/m2. Inclusion criteria for individuals without T2D; no diagnosis of T2D, male gender, age > 40 years, and BMI < 35 kg/m2. Exclusion criteria for all participants; trombocyte count < 100, treatment with anticoagulants except acetylic acids, renal impairment (eGFR <50 ml/min), bone metabolic disease, vitamin D insufficiency, treatment with antiosteoporotic agents or systemic glucocorticoids, and tetracycline allergy.

3.11 Methods Fasting morning blood samples will be collected. The participants will undergo a whole body dual energy x-ray absorptiometry (DXA) to investigate body composition (lean and fat mass) and a Jamshidi bone marrow biopsy in which two pieces of bone tissue is collected for measurement of bone turnover and AGES.

3.12. Bone tissue biopsy Before the bone tissue sampling, the bone tissue will be labelled twice by administration of tetracycline. Tetracykline is incorporated in newly formed bone as bands that are visible in a microscope. A histomorphometric analysis is conducted on the bone tissue sample to investigate the indices of bone turnover.

3.13 Measurement of biomarkers From the bone marrow and plasma/serum samples the following is measured Bone resorption markers: CTX and TRAP5b. Bone formation markers: P1NP, Osteocalcin, and Bone specific alkaline phosphatase.

Bone signaling markers: Osteoprotegerin, RANKL, Sclerostin and parathyroid hormone.

3.14. Analysis of the whole body DXA The whole body DXA measures BMD and lean and fat mass. 3.15 Measurement of AGEs Blood serum and bone marrow serum levels of AGEs are measured. For each participant, one bone tissue biopsy is pulverized, and the level of AGEs in the bone tissue estimated by Fourier Transformed Infrared Spectroscopy (FTIR) in collaboration with the Interdisciplinary Nanoscience Center, Aarhus University. Skin autofluorescence will be applied to non-invasively measure levels of AGEs in the skin.

3.16 Statistics Students t-tests will be used to compare levels of bone turnover markers and AGEs between individuals with and without T2D. Bland Altman plots will be used to analyze agreement between measurement of the bone turnover markers and AGEs at the different tissue compartments. Adjustment will be performed using logistic or linear regression dependent on data distribution.

3.1.7 Power calculation The power calculation is based on the bone formation marker, osteocalcin. Plasma osteocalcin levels were in a previous study 14,4 +/- 5,3 ug/l (mean+/-SD).

It is expected that tere will be a 30% lower level of osteocalcin in individuals with T2D compared to individuals without T2D. Based on the above assumptions, the probability of a type 1 error of 0.05, the probability of a type II error of 0.8, and that two marrow aspirations in each group will fail, 26 individuals should be included in each group in order to detect a difference.

3.l.8 Approval The study is approved at the Regional Ethics Committee, Region Midtjylland: 1-10-72-214-21.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for individuals with T2D;

* physician diagnosed T2D,
* diabetes duration ≥5 years,
* HbA1c ≥ 48 mmol/mol through the last 2 years
* male gender,
* age > 40 years
* BMI < 35 kg/m2

Inclusion criteria for individuals without T2D;

* no diagnosis of T2D
* male gender,
* age > 40 years
* BMI < 35 kg/m2

Exclusion Criteria:

* trombocyte count < 100
* treatment with anticoagulants except acetylic acids,
* renal impairment (eGFR <50 ml/min),
* bone metabolic disease
* vitamin D insufficiency
* treatment with antiosteoporotic agents
* Treatment with systemic glucocorticoids
* Tetracycline allergy.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 26 individials with type 2 diabetes and 26 controls without type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of Osteocalcin | 2 years
  Circulating bone turnover marker

SECONDARY OUTCOMES:
Plasma concentration of CTX | 2 years
  Circulating bone turnover marker
Plasma concentration of P1NP | 2 years
  Circulating bone turnover marker
Plasma concentration of Sclerostin | 2 years
  Circulating bone turnover marker
Bone marrow serum concentration of P1NP | 2 years
  Circulating bone turnover marker
Bone marrow serum concentration of CTX | 2 years
  Circulating bone turnover marker
Bone marrow serum concentration of Osteocalcin | 2 years
  Circulating bone turnover marker
Bone marrow serum concentration of Sclerostin | 2 years
  Circulating bone turnover marker
serum concentration of penstosidine | 2 years
  Advanced glycation endproduct
bone marrow serum concentration of pentosidine | 2 years
  Advanced glycation endproduct
Bone formation rate in bone tissue | 2 years
  Bone turnover in bone based on histomorphometric analysis
Advanced glycation endproductsproducts in bone | 2 years
  Raman spectroscopy to determine levels of Advanced glycation endproducts in bone tissue
Strenght measure of bone | 2 years
  Nano-indentation of the bone
trabecular separation distance | 2 years
  bone structure measure provided by x-ray nano-CT

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to GPRD it may not be possible to share IPD.